CLINICAL TRIAL: NCT07205211
Title: Attention Deficit Hyperactivity Disorder (ADHD) Symptoms in Children With Epilepsy
Brief Title: Prevalence of ADHD in Children With Epilepsy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Menna Allah Abdelrazek Ali Gad Kassab, Principal investigator, Assiut University
Other Study IDs: ADHD in pediatric epilepsy
Record Dates: First submitted 2025-09-13; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: ADHD; Epilepsy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To Determine the prevalence of ADHD symptoms in children with epilepsy, And find out the possible risk factors of ADHD in such patients and it's effect on prognosis of the disease

DETAILED DESCRIPTION:
Epilepsy may be defined as the recurrence of apparently spontaneous seizures and can be a pervasive condition in which the seizures are just one expression Epileptic seizures are transient clinical events resulting from atypical and excessive activity of more or less widespread population of cerebral neurons Epilepsy is a heterogeneous disorder that consists of clinical syndromes, characterized by different types of seizures, and underlying aetiologies . It is the most common pediatric neurological disorder with prevalence estimates of 0.5-1% of all children from birth to 16 years .

Attention deficit/hyperactivity disorder (ADHD) is a common brain disorder with onset in early childhood,due to structural and functional abnormalities in widespread, but specific areas of the brain . ADHD is a frequent co morbidity experienced by children with epilepsy, has a negative impact on their quality of life,and represents a significant risk factor for academic underachievement.

ADHD has been reported in epilepsy since the Fifties of the 20th century .More recently a high association between the two disorders, with an increasing evidence of a bidirectional relationship, has been postulated . Several factors may contribute to this comorbidity, including the underlying brain pathology, the chronic effects of seizures and of the epileptiform EEG discharges, and the effects of antiepileptic drugs. Symptoms of ADHD are more common in some specific types of epilepsies, such as frontal lobe epilepsy, childhood absence epilepsy and Rolandic epilepsy, and may antedate seizure onset in a significant proportion of cases.

Attention problems are frequently reported in children with intractable symptomatic epilepsy, as well as in idiopathic epilepsies . Patients who have generalized epilepsies are more frequently reported to have attentional difficulties than patients suffering from partial seizures. Furthermore, certain epilepsy syndromes may predispose to ADHD-like behavior .ADHD is a prevalent co morbidity of new onset idiopathic epilepsy, associated with a series of cognitive and behavioral complications that antedate epilepsy onset in a significant proportion of cases, and appear related to neurodevelopmental abnormalities in brain structures . The presence of ADHD symptoms at the time of epilepsy onset is a major marker of abnormal cognitive development The mechanisms underlying attention deficits are still unknown and appear to be different between focal and generalized epilepsies. In the clinical practice, this association may represent a challenge for child neurologists since antiepileptic therapy and drugs used to treat ADHD may aggravate the clinical picture of each other .-Treatment with psychotropic drugs can be initiated safely in most children with epilepsy and ADHD symptoms.

Previous studies show that Children with epilepsy have more attention problems as compared with healthy controls. ADHD in childhood epilepsy is associated with male sex, younger age, early first onset age, high frequency of epileptic seizures, and multiple AEDs

ELIGIBILITY:
Inclusion Criteria:

All children above the age of 3 years who have any type of epilepsy and are seen in the neurology unit in Assiut University Children's Hospital.

Exclusion Criteria:

Children below 3 years of age. Children with ADHD who do not have epilepsy.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consists of children above 3 years with epilepsy and develop symptoms of ADHD or even have ADHD before diagnosis of epilepsy And compared with those with epilepsy but don't develop ADHD to determine the prevalence,risk factor And the prognosis. participants will be recruited from pediatric neurology unit & neurology outpatiend clinic in Assuit University Children's Hospital
Sampling Method: Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in ADHD Symptom Total Score (ADHD-SC4) | 12 weeks
  The primary outcome will be the change from baseline in the total symptom score, as measured by the ADHD Symptom Checklist-4 Scale (ADHD-SC4), a validated parent-completed rating scale. Efficacy will be determined by a statistically significant reduction in the total score from baseline to the final 12-week assessment compared to control.

SECONDARY OUTCOMES:
Change from Baseline in Quality of Life Total Score (PedsQL™ 4.0 Generic Core Scales) | 12 weeks
  The change from baseline to the final 12-week assessment in the overall Total Score from the Pediatric Quality of Life Inventory™ 4.0 Generic Core Scales (PedsQL). The PedsQL is a validated, patient- and parent-reported scale that assesses daily functioning, social relationships, and emotional health. The total score will be used as the primary QoL metric.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kanner AM. The use of psychotropic drugs in epilepsy: what every neurologist should know. Semin Neurol. 2008 Jul;28(3):379-88. doi: 10.1055/s-2008-1079342. Epub 2008 Jul 24. PMID 18777484
- [Result] Caplan R, Siddarth P, Stahl L, Lanphier E, Vona P, Gurbani S, Koh S, Sankar R, Shields WD. Childhood absence epilepsy: behavioral, cognitive, and linguistic comorbidities. Epilepsia. 2008 Nov;49(11):1838-46. doi: 10.1111/j.1528-1167.2008.01680.x. Epub 2008 Jun 13. PMID 18557780
- [Result] Steer CR. Managing attention deficit/hyperactivity disorder: unmet needs and future directions. Arch Dis Child. 2005 Feb;90 Suppl 1(Suppl 1):i19-25. doi: 10.1136/adc.2004.059352. PMID 15665152
- [Result] OUNSTED C. The hyperkinetic syndrome in epileptic children. Lancet. 1955 Aug 13;269(6885):303-11. doi: 10.1016/s0140-6736(55)92304-7. No abstract available. PMID 13243723
- [Result] Davies S, Heyman I, Goodman R. A population survey of mental health problems in children with epilepsy. Dev Med Child Neurol. 2003 May;45(5):292-5. doi: 10.1017/s0012162203000550. PMID 12729141
- [Result] Hermann B, Jones J, Dabbs K, Allen CA, Sheth R, Fine J, McMillan A, Seidenberg M. The frequency, complications and aetiology of ADHD in new onset paediatric epilepsy. Brain. 2007 Dec;130(Pt 12):3135-48. doi: 10.1093/brain/awm227. Epub 2007 Oct 18. PMID 17947336
- [Result] Schubert R. Attention deficit disorder and epilepsy. Pediatr Neurol. 2005 Jan;32(1):1-10. doi: 10.1016/j.pediatrneurol.2004.06.007. PMID 15607597
- [Result] Dunn DW, Kronenberger WG. Childhood epilepsy, attention problems, and ADHD: review and practical considerations. Semin Pediatr Neurol. 2005 Dec;12(4):222-8. doi: 10.1016/j.spen.2005.12.004. PMID 16780293
- [Result] Torres AR, Whitney J, Gonzalez-Heydrich J. Attention-deficit/hyperactivity disorder in pediatric patients with epilepsy: review of pharmacological treatment. Epilepsy Behav. 2008 Feb;12(2):217-33. doi: 10.1016/j.yebeh.2007.08.001. Epub 2007 Dec 11. PMID 18065271